CLINICAL TRIAL: NCT05909241
Title: A Multicenter, Open-label, Single-arm, Dose Escalation and Expansion Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of BA1202 in Patients With Advanced Solid Tumors
Brief Title: A Study of BA1202 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Boan Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BA1202/CT-CHN-101
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BA1202 (Experimental): BA1202 is a bispecific antibody targeting CEA and CD3.
  Interventions: Drug: BA1202

INTERVENTIONS:
Drug: BA1202 — BA1202 will be administered intravenously (IV) once every 3 weeks (Q3W) until confirmed progression, death, unaccepted toxicity, initiation of other antitumor therapies, or any other conditions requiring treatment discontinuation, and the duration of administration was no more than 2 years.
  Part A: Patients will receive one of the following dosages of BA1202: 0.016mg, 0.08mg, 0.4mg, 1.6mg, 6.4mg, 19mg, 38mg, 56mg.
  Part B: Based on the data of part A, one or two dose levels will be discussed for further evaluation in part B.

SUMMARY:
This is a multicenter, open-label, single-arm phase I study in patients with advanced solid tumors which consists of a dose escalation part (Part A) and a dose extension part (Part B).

Part A aims to evaluate the safety and tolerability of BA1202, and determine the MTD. Part B will also evaluate the preliminary efficacy of BA1202.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily sign an IRB-approved informed consent form, and are willing to abide by the restrictions of the study.
* Part A: Patients with histologically and/or cytologically confirmed advanced and/or metastatic solid tumors who have progressed on Standard-Of-Care (SOC), are intolerant to SOC, or have no SOC.
* Part B: Patients with histologically and/or cytologically confirmed colorectal cancer, non-small cell lung cancer, pancreatic cancer, gastric cancer, who have progressed on Standard-Of-Care (SOC), are intolerant to SOC, or have no SOC.（Specific cohort will be determined after data of dose escalation phase is obtained）
* Part B: High expression of CEACAM5 (defined as ≥ 20% of tumor cells with IHC 2+ and/or 3+).
* Life expectancy of at least 3 months.
* At least one evaluable lesion in Part A and at least one measurable lesion in Part B according to RECIST v1.1.
* ECOG score of < 2.
* Absolute neutrophil count ≥ 1.5 x 10^9/L, platelet count ≥ 100 x 10^9/L, hemoglobin ≥ 90 g/L.
* Total bilirubin ≤ 1.5×ULN, ALT and AST ≤ 2.5×ULN (or ≤ 5.0×ULN for patients with liver metastases).
* Serum creatinine ≤ 1.5×ULN, or creatinine clearance ≥50 mL/min.
* International normalized ratio (INR) prothrombin time (PT) ≤1.5×ULN, activated partial thromboplastin time (APTT) ≤1.5×ULN.
* Blood pregnancy test results were negative for female patients with fertility potential. Patients with fertility potential must agree to use a reliable method of contraception with their sexual partners during the study period and at least 6 months after the last administration.

Exclusion Criteria:

* Other malignancies within 5 years prior to screening (other than cured stage Ib or lower cervical cancer, non-invasive basal cell or squamous cell skin cancer).
* Has a persistent or active infection that requires intravenous treatment.
* History of severe cardiovascular and cerebrovascular disease.
* Patients with autoimmune diseases requiring drug control or at risk of recurrence of autoimmune diseases.
* Received any radiotherapy (other than palliative radiotherapy for bone metastases), chemotherapy, targeted therapy, immunotherapy, cell therapy, or other investigational anticancer agents within 4 weeks prior to first dose of BA1202, unless chemotherapy or targeted therapy is less than 4 weeks after first dose but has eluted ≥5 half-lives.
* Have received any previous CEA targeting therapy, including but not limited to monoclonal antibodies, bisspecific antibodies, antibody-coupled drugs (ADCs), chimeric antigen receptor T cells (CAR-T), etc.
* A history of allergy to BA1202 or any component of Obinutuzumab, or to other monoclonal antibodies.
* Women are planning to become pregnant or are pregnant or breastfeeding.
* Other conditions considered unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment, up to 2 years.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of BA1202 | Cycle 1: Day 1, 2, 3, 5, 8, 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 4: Day 1, 2, 3, 5, 8, 15; Cycle 5 Day 1; Cycle 6 Day 1. (Each cycle is 21 days.)
Area under the curve (AUC) of BA1202 | Cycle 1: Day 1, 2, 3, 5, 8, 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 4: Day 1, 2, 3, 5, 8, 15; Cycle 5 Day 1; Cycle 6 Day 1. (Each cycle is 21 days.)
Minimum Concentration (Cmin) of BA1202 | Cycle 1: Day 1, 2, 3, 5, 8, 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 4: Day 1, 2, 3, 5, 8, 15; Cycle 5 Day 1; Cycle 6 Day 1. (Each cycle is 21 days.)
Time of maximum concentration (Tmax) of BA1202 | Cycle 1: Day 1, 2, 3, 5, 8, 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 4: Day 1, 2, 3, 5, 8, 15; Cycle 5 Day 1; Cycle 6 Day 1. (Each cycle is 21 days.)
Objective Response Rate (ORR) | up to 2 years
Disease Control Rate (DCR) | up to 2 years
Duration of Response (DOR) | up to 2 years
Overall Survival (OS) | up to 2 years
Progression-Free Survival (PFS) | up to 2 years
Proportion of subjects with positive anti-drug antibody (ADA) and neutralizing antibody (Nab) | Cycle 1: Day 1, 15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 4 Day 1; Cycle 5 Day 1; Cycle 6 Day 1; EOT (end of treatment) visit. (Each cycle is 21 days.)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China